CLINICAL TRIAL: NCT00187850
Title: The CAP-2 Trial: Effect of Direct Pulp Capping Versus Partial Pulpotomy on CAP-1 Patients: A Randomised, Patient - and Observer-Blinded Multicenter Trial
Brief Title: The CAP-2 Trial: Effect of Direct Pulp Capping Versus Partial Pulpotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: National Health Insurance foundation (Unknown); Dan Dental A/S (Industry); University of Aarhus (Other); Göteborg University (Other); Huddinge Faculty,Stockholm,Sweden (Unknown); Uppsala FolkTandvård,Sweden (Other); Malmö Dental school,Sweden (Unknown)
Responsible Party: Principal Investigator, Lars Bjørndal, PhD, Dr.Odont, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10002
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Dental Pulp Exposure
Keywords: Pulp capping; partial pulpotomy; Exposure of the pulp
MeSH Terms: conditions — Dental Pulp Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PP (Experimental): Partial pulpotomy
  Interventions: Procedure: PP
- DPC (Other): Direct pulp capping
  Interventions: Procedure: DPC

INTERVENTIONS:
Procedure: PP — Partial pulpotomy
  Other Names: cvek´s pulpotomy
  Arms: PP
Procedure: DPC — Direct pulp capping
  Arms: DPC

SUMMARY:
CAP-2 Trial

Background: This trial is being done in conjunction with an ongoing clinical trial investigating stepwise excavation versus final excavation on deep caries lesions (The CAP-1 trial). The investigators lack systematic knowledge concerning the treatment of the exposed pulp and whether the capping of a pulp represents the same outcome as the partial removal of an additional 1-1.5 mm of the pulp tissue (partial pulpotomy).

Aim: The aim of the CAP-2 trial is in a randomised clinical trial to investigate the effect of direct pulp capping versus partial pulpotomy in patients who, from the beginning, have received either a final excavation or a stepwise excavation and where this intervention has led to the exposure of a vital pulp and/or the patient has not gained relief from tooth pain after excavation and placement of a temporary restoration.

Patients: Patients include consecutive patients with deep caries who have been participating in the CAP-1 trial, where the pulp exposure to a bleeding pulp is present and/or pain relief has not been obtained.

Design: The CAP-2 trial is a randomised patient- and observer-blinded multicenter trial, with two parallel intervention groups. Patients who fulfill the inclusion criteria will be centrally bloc-randomised in the Copenhagen Trial Unit, Copenhagen DK, and stratified by age and pain. The allocation ratio is 1:1.

The Interventions and Products: Patients are allocated for direct pulp capping or partial pulpotomy. The patients will not be informed about the results of the randomisation, i.e. the type of intervention. In both groups the patient receives a calcium hydroxide seal covering the exposure and a glass ionomer restoration. The final resin restoration is placed following 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Persons participating in the CAP-1 trial, who have received a pulp exposure due to treatment or due to absence of pain relief.

Exclusion Criteria:

* The CAP-1-treated tooth has ongoing unbearable pain and/or disturbed night sleep.
* Visible pus from the pulp.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-02; Primary Completion 2007-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The survival of the tooth with vital pulp and without apical radiolucency. The x-ray evaluation and the clinical sensibility test are carried out by a blinded observer. | 1 year after inclusion in the CAP-2

SECONDARY OUTCOMES:
Gain of pain relief | after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bjørndal, Ph.D., Study Director — University of Copenhagen
Locations (1):
- Copenhagen University, Copenhagen, Copenhagen N, Denmark

REFERENCES:
- [Background] Bjorndal L, Reit C, Bruun G, Markvart M, Kjaeldgaard M, Nasman P, Thordrup M, Dige I, Nyvad B, Fransson H, Lager A, Ericson D, Petersson K, Olsson J, Santimano EM, Wennstrom A, Winkel P, Gluud C. Treatment of deep caries lesions in adults: randomized clinical trials comparing stepwise vs. direct complete excavation, and direct pulp capping vs. partial pulpotomy. Eur J Oral Sci. 2010 Jun;118(3):290-7. doi: 10.1111/j.1600-0722.2010.00731.x. PMID 20572864
- [Derived] Bjorndal L, Fransson H, Bruun G, Markvart M, Kjaeldgaard M, Nasman P, Hedenbjork-Lager A, Dige I, Thordrup M. Randomized Clinical Trials on Deep Carious Lesions: 5-Year Follow-up. J Dent Res. 2017 Jul;96(7):747-753. doi: 10.1177/0022034517702620. Epub 2017 Apr 14. PMID 28410008